CLINICAL TRIAL: NCT02073370
Title: Clinical Evaluation, Biomarkers and Metabolomics of Sarcopenia in Frail Older Adults at Ambulatory Clinics
Acronym: EC0991002-E
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Health Research Institutes, Taiwan (Other); National Taiwan University (Other)
Responsible Party: Sponsor
Other Study IDs: 201010021R; EC0991002-E (Registry Identifier: NHRI EC0991002-E)
Record Dates: First submitted 2011-08-30; First posted 2014-02-27 (Estimated); Last update posted 2014-02-27 (Estimated); Status verified 2014-02

CONDITIONS: Frailty; Sarcopenia
MeSH Terms: conditions — Frailty; Sarcopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- health subjects; outpatients aged over 65: The research subjects will be culled from outpatients aged over 65 at NTUH; 1000 Taiwanese subjects aged 20-40 equally divided in both genders will be recruited in order to establish the norm of Taiwanese's skeletal muscle index.

SUMMARY:
Sarcopenia related mobility dysfunction was a preventable presentation in transitional variation of frailty. However, the definition, associated risk factors, clinical course and outcome of sarcopenia in Taiwanese older adults are still under-clarified and need for further study.

ELIGIBILITY:
Inclusion Criteria:

* functional decline in recent one year
* cognitive impairment
* depressive symptom
* mobility impairment
* fall in recent one year
* eating or feeding problems
* weight loss
* co-morbid conditions≧5
* tracking by different physician ≧3 in recent half year
* poly-pharmacy≧8 in recent 3 months
* hospitalization ≧1 in recent one year
* emergency visits≧2 in recent one year
* aged ≧ 80.

Exclusion Criteria:

* non-ambulatory (bed-ridden) patients
* long-term residents at nursing homes
* patients with a life expectancy shorter than six months
* impairment in vision, hearing, or communicative ability, making convenience of clinical evaluation during the study period impossible.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Healthy subjects One thousand Taiwanese subjects aged 20-40 will be recruited equally divided in both genders. Exclusion criteria includes (1) morbid obesity (BMI over 35) ; (2) long term use of body composition modified medications, like steroid, medications for endocrine diseases (hyperthyroidism, diabetes) and autoimmune diseases; (3) energy consumption diseases, such as cancer, organ failure; (4) pregnant women.
  Patient enrollment The research subjects will be culled from outpatients aged over 65 at NTUH.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2011-01; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Domestic operation tool of sarcopenia for older adults | Baseline
  Young health adults are recruited for measurement of body composition using bio impedance analysis in order to establish the norm of skeletal muscle index

SECONDARY OUTCOMES:
Change from baseline in body composition during aging | up to 2 years
  Using anthropometric measurements, and bio impedance analysis, the change in body composition are measured in the recruited older adults

OTHER OUTCOMES:
Compare metabolomics profiles in sarcopenic older adults and non-sarcopenic older adults | up to 2 years
  Using the blood specimen, the metabolomics platform are set up to explore the new bio markers of sarcopenia in older adults
The prognosis of sarcopenia in the older adults | up to 2 years
  The adverse health outcomes, including hospitalization, emergency visits, or fall events, are recorded every 3 months in order to examine the prognosis of sarcopenia in the elderly

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Yu Chen, MD, Principal Investigator — National Tiwan University, College of Medicine
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan